CLINICAL TRIAL: NCT01778751
Title: Advanced Comprehensive Diabetes Care for Veterans With Poorly-Controlled Diabetes
Acronym: ACDC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RRP 12-458
Record Dates: First submitted 2013-01-18; First posted 2013-01-29 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes
Keywords: Self-Management Support; Depression; Home Telehealth
MeSH Terms: conditions — Diabetes Mellitus; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Veterans will receive diabetes educational materials and management per their primary provider
- Intervention (Experimental): Veterans randomized to the intervention arm will be enrolled in the HT program, provided with standard telemonitoring equipment by HT nursing staff (current HT practice at DVAMC is use of the Health Buddy 3 device for patients with landline phones and the Cardiocom Interactive Voice Response System for patients with cell phones), and will receive the study intervention for 6 months. Veterans without depressive symptoms on baseline PHQ-9 assessment (PHQ-9 < 10) will not initially be entered into the depressive symptom management component of the intervention, but will be monitored for new symptoms throughout the intervention.
  Interventions: Behavioral: Home Telehealth with Behavioral Education Component

INTERVENTIONS:
Behavioral: Home Telehealth with Behavioral Education Component — The primary effectiveness outcome for this study will be hemoglobin A1c. Secondary effectiveness outcomes will include measures of diabetes self-care, self-reported medication adherence, and depressive symptoms.
  Arms: Intervention

SUMMARY:
This study will determine whether Home Telehealth-based implementation of an evidence-based intervention targeting Veterans with persistent poorly-controlled diabetes can improve hemoglobin A1c, patient self-management, and comorbid depressive symptoms in this high-risk, high-cost population. If effective, this intervention (Advanced Comprehensive Diabetes Care) offers a feasible, sustainable, and generalizable approach to managing Veterans with persistent poorly-controlled diabetes, which can be implemented using only existing Home Telehealth services.

DETAILED DESCRIPTION:
Background: Although efforts by VA providers and researchers have improved diabetes care quality for Veterans, individuals with persistent poorly-controlled diabetes mellitus (type 1 or type 2 diabetes with hemoglobin A1c >9.0% for > 1 year despite receipt of medical care) have proven refractory to these widespread improvements, and remain at high risk for complications and accrued costs. Prior research has illustrated that medication regimen complexity, suboptimal self-care, and comorbid depressive symptoms interact to perpetuate suboptimal control among individuals with PPDM. Current models of clinic-based diabetes care do not meet these Veterans' needs. Without the implementation of care delivery strategies that target this population's unique barriers to improved diabetes control, these Veterans will continue to be left behind by progress in diabetes management throughout VA, and will remain at high risk for complications and high costs. We propose using existing local Home Telehealth services to implement Advanced Comprehensive Diabetes Care, a patient-centered, evidence-based intervention combining medication management, self-care behavior support, and depressive symptom management to Veterans with PPDM.

Objectives: The specific aims of this RRP are to: 1) evaluate the effectiveness of the Advanced Comprehensive Diabetes Care among Veterans with persistent poorly-controlled diabetes; 2) utilize a mixed method formative evaluation to assess our main implementation strategy, the use of existing Home Telehealth services to administer the intervention; and 3) generate data we will use to refine local intervention implementation and inform the development of an SDP proposal evaluating broader implementation of the Advanced Comprehensive Diabetes Care intervention.

Methods: We propose a pilot Effectiveness-Implementation Hybrid trial to study the Advanced Comprehensive Diabetes Care intervention in Veterans with persistent poorly-controlled diabetes. After baseline evaluation, 50 Veterans will be randomly assigned into intervention (n = 25) or control groups (n = 25). Veterans randomized to the intervention will be enrolled in the Home Telehealth program at Durham VAMC and will receive the study intervention (telehealth-based medication management, self-care behavior support, and depressive symptom management) for 6 months. Intervention-group Veterans with no depression on baseline assessment will not initially receive the depressive symptom management component, but will be monitored for new symptoms throughout the study. Veterans randomized to the control arm will receive diabetes educational materials and management per their primary provider. The primary effectiveness outcome for this study will be hemoglobin A1c. Secondary effectiveness outcomes will include measures of diabetes self-care, self-reported medication adherence, and depressive symptoms. This RRP will also include a mixed method formative evaluation to qualitatively and quantitatively assess patient-level, provider-level, and organizational barriers and facilitators influencing intervention implementation. Formative evaluation data will be analyzed during the study to consider whether adjustments to the intervention or its implementation may be indicated, and findings will also be used to inform future implementation efforts.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with type 2 diabetes managed for > 1 year at an eligible site (Durham, Raleigh, Greenville, or Morehead City) will be eligible for enrollment.
* We will identify Veterans with PPDM (defined as the presence of at least 2 A1c values of > 9.0% during the past year with no readings of < 9.0% despite ongoing medical care) by reviewing electronic medical records and soliciting referrals from primary physicians.

Exclusion Criteria:

* Exclusion criteria will include lack of telephone access or severe hearing/ speech impairment that would limit:

  * telephone interaction
  * metastatic cancer
  * active psychosis documented in medical record
  * active alcohol or substance abuse
  * diagnosis of dementia
  * known pregnancy (patients becoming pregnant during the study will be withdrawn and referred to appropriate services)
  * documented seizure history
  * documented history of severe complications of hypoglycemia (such as coma or seizure)
  * documented refusal or inability to perform self-monitoring of blood glucose
  * ongoing use of warfarin with prior history of major bleeding event
* Due to challenges with dose adjustment by phone, Veterans on continuous subcutaneous insulin infusion (insulin pumps) will not be eligible for this study.

  * Due to challenges with regulations regarding testing supplies pts will need to be taking insulin (a few patients had enrolled prior to this change.).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Crowley, MD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Derived] Crowley MJ, Edelman D, McAndrew AT, Kistler S, Danus S, Webb JA, Zanga J, Sanders LL, Coffman CJ, Jackson GL, Bosworth HB. Practical Telemedicine for Veterans with Persistently Poor Diabetes Control: A Randomized Pilot Trial. Telemed J E Health. 2016 May;22(5):376-84. doi: 10.1089/tmj.2015.0145. Epub 2015 Nov 5. PMID 26540163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred December 2013-May 2014 at the Durham VA Medical Center outpatient primary care clinics.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 25 | 25
Completed | 23 | 23
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Transfered care | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.2) | 60.2 (8.4) | 59.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 25 | 23 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 8 | 13 | 21
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Control
Description: Hemoglobin A1c as measured at baseline, 3m, 6m
Time Frame: Baseline, 3months, 6months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Control | Intervention
Number analyzed (Participants) | 25 | 25
percentage of glycosylated hemoglobin
  Baseline | 10.7 (1.6) | 10.2 (1.4)
  3 Months | 10.3 (1.8) | 9.1 (1.3)
  6 months | 10.4 (1.6) | 9.1 (2.1)
Statistical Analysis 1: Comparison: Control vs Intervention; Comparison at 3 months; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis; Mean Difference (Net) = -1.0, 95% CI 2-sided [-1.7 to -0.2]
Statistical Analysis 2: Comparison: Control vs Intervention; Comparison at 6 months; Test type: Superiority or Other; p = 0.050, Mixed Models Analysis; Mean Difference (Net) = -1.0, 95% CI 2-sided [-2.0 to -0.0]

2. Secondary Outcome: Diabetes Self Care
Description: Self-Care Inventory-revised as measured at baseline, 3 months, 6 months
Time Frame: Baseline, 3m, 6m
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline | 49.8 (9.6) | 52.3 (14.8)
  3 months | 53.7 (10.9) | 58.2 (14.6)
  6 months | 52.6 (12.6) | 61.1 (14.0)
Statistical Analysis 1: Comparison: Control vs Intervention; Comparison at 3 months, Scale is 0-100 where a higher score is a better outcome; Test type: Superiority or Other; p = 0.303, Mixed Models Analysis; Mean Difference (Net) = 2.9, 95% CI 2-sided [-2.7 to 8.4]
Statistical Analysis 2: Comparison: Control vs Intervention; Comparison at 6 months, Scale is 0-100 where a higher score is a better outcome; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis; Mean Difference (Net) = 7.7, 95% CI 2-sided [0.9 to 14.4]

3. Secondary Outcome: Self-reported Medication Adherence
Description: Change in Self-Reported Medication- Taking Scale as measured at baseline, 3 months, 6 months
Time Frame: Baseline, 3m, 6m
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 25 | 25
participants
  Baseline | 17 | 15
  3 months | 11 | 9
  6 months | 9 | 8
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.830, Generalized estimating equation (GEE); Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.35 to 2.34]
Statistical Analysis 2: Comparison: Control vs Intervention; Comparison at 6 months; Test type: Superiority or Other; p = 0.970, Generalized Estimating Equation (GEE); Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.33 to 3.19]

4. Secondary Outcome: Depressive Symptoms
Description: Change in Patient Health Questionnaire as measured at Baseline, 3 months, 6 months
Time Frame: Baseline, 3m, 6m
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline | 7.3 (5.5) | 6.9 (5.6)
  3 months | 6.6 (5.1) | 5.5 (6.3)
  6 months | 5.9 (4.7) | 6.7 (6.2)
Statistical Analysis 1: Comparison: Control vs Intervention; Comparison at 3 months. Scale is 0-27 where a lower score is a better outcome, values were dichotomized to indicate whether or not the patient was depressed; Test type: Superiority or Other; p = 0.428, Mixed Models Analysis; Mean Difference (Net) = -0.9, 95% CI 2-sided [-3.3 to 1.4]
Statistical Analysis 2: Comparison: Control vs Intervention; Comparison at 6 months. Scale is 0-27 where a lower score is a better outcome, values were dichotomized to indicate whether or not the patient was depressed; Test type: Superiority or Other; p = 0.397, Mixed Models Analysis; Mean Difference (Net) = 1.1, 95% CI 2-sided [-1.4 to 3.6]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at 3 and 6 months for all participants. Participants randomized to the intervention arm were monitored on a more frequent basis during the intervention telephone contacts.
Description: Patients were asked about recent health events and the medical records were reviewed at each follow-up assessment (3&6mths). Participants participating in the intervention were monitored via the home telehealth equipment and intervention telephone contacts.
Arm/Group | Control | Intervention
Serious Adverse Events (participants affected / at risk) | 4/25 | 3/25
Other Adverse Events (participants affected / at risk) | 12/25 | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=25) | Intervention (N=25)
Hospitalization (Cardiac disorders) | 1 (1) | 1 (1)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hospitalization (General disorders) | 0 (0) | 1 (1)
Hospitalization (Renal and urinary disorders) | 0 (0) | 1 (1)
Outpatient Diagnosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0)
Psychiatric Disorder (Psychiatric disorders) | 1 (1) | 0 (0) — Emergency Room Visit
Hypoglycemia Requiring Asssistance (Investigations) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=25) | Intervention (N=25)
Biopsy (Endocrine disorders) | 0 (0) | 1 (1) — Thyroid nodule
Biopsy (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) — Skin biopsy
Ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Emergency Room Visit
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1) — Emergency Room Visit
Eye pain (Eye disorders) | 1 (1) | 0 (0) — Emergency Room Visit
Emergency Room Visit (General disorders) | 6 (12) | 7 (9) — We collected adverse events by organ system and categorized them using the Emergency Room distinction. Affected patients may have visited the ER for a range of conditions (for instance pain, cuts, medication refills, etc)
Emergency Room Visit (Infections and infestations) | 1 (1) | 3 (3) — We collected adverse events by organ system and categorized them using the Emergency Room distinction. Affected patients may have visited the ER for a range of conditions (for instance coughs, illnesses, etc)
Emergency Room Visit (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) — We collected adverse events by organ system and categorized them using the Emergency Room distinction. Affected patients may have visited the ER for a range of conditions (for instance pain, etc)
Psychiatric Disorder (Psychiatric disorders) | 1 (1) | 0 (0) — Emergency Room Visit
Emergency Room Visit (Renal and urinary disorders) | 1 (1) | 2 (2) — We collected adverse events by organ system and categorized them using the Emergency Room distinction. Affected patients may have visited the ER for a range of conditions (for instance pain associated with stones, etc)
Emergency Room Visit (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — We collected adverse events by organ system and categorized them using the Emergency Room distinction. Affected patients may have visited the ER for a range of conditions (for instance cough, etc)
cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Emergency Room Visit
Emergency Room Visit (Vascular disorders) | 1 (1) | 1 (1) — We collected adverse events by organ system and categorized them using the Emergency Room distinction. Affected patients may have visited the ER for a range of conditions (for instance swelling, bleeding, etc)
Planned Surgery and Proceedures (Surgical and medical procedures) | 1 (1) | 2 (3)
# Pts with >5 BG Values <70 mg/dL from 1st encounter to end of study (Investigations) | 0 (0) | 3 (3) — Telehealth reported data (intervention group only)-

LIMITATIONS AND CAVEATS:
* Single-center pilot study
* Small, male Veteran population with type 2 diabetes
* Uses VA-specific infrastructure, findings may not translate to other settings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes